CLINICAL TRIAL: NCT00582179
Title: Vacuum Assisted Closure as a Treatment For Draining Hematomas (Vacuum Assisted Closure in the Management of Traumatic Extremity Wounds)
Brief Title: Vacuum Assisted Closure as a Treatment for Draining Hematomas
Acronym: VAC-DH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F010316005
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Draining Hematoma
Keywords: Draining Hematoma; Vacuum Assisted Closure (VAC); Negative Pressure Wound Therapy (NPWT); Draining Hematoma following orthopaedic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, A (Active Comparator): Group A patients will be treated with a pressure dressing and observation.
  Interventions: Procedure: Standard Pressure Dressing
- 2, B (Active Comparator): Group B patients will be treated with a Vacuum Assisted Closure device (VAC).
  Interventions: Device: VAC

INTERVENTIONS:
Procedure: Standard Pressure Dressing — If hematoma still draining at 5 days post surgery, patients who randomize to Group A will have a standard pressure dressing applied and checked every 24-48 hours for continued draining. If still draining at 10 days post surgery, patient is at end point of study and must return to OR for Irrigation and Debridement of the wound. If infection occurs, patient is at end point of study and must return to OR for I&D.
  Arms: 1, A
Device: VAC — If hematoma still draining at 5 days post surgery, patients who randomize to Group B will have a VAC negative pressure device applied and checked every 24-48 hours for continued draining. If still draining at 10 days post surgery, patient is at end point of study and must return to OR for Irrigation and Debridement of the wound. If infection occurs, patient is at end point of study and must return to OR for I&D.
  Other Names: Vacuum Assisted Closure device, Kinetics Concepts, Inc.
  Arms: 2, B

SUMMARY:
This project is designed as a prospective, randomized, comparative study evaluating the use of a negative pressure vacuum device in treating draining hematomas following traumatic injury.

DETAILED DESCRIPTION:
Application of the VAC device may significantly decrease the incidence of draining hematomas that require surgical irrigation and debridement. The aim of this project is to perform a prospective, randomized study evaluating the VAC negative pressure device as a treatment for draining hematomas. We will also analyze the cost of treating a hematoma with a VAC compared with currently employed treatments. Additionally, we will document the incidence of infection of the hematoma with and without use of the VAC device.

Patients who have a draining hematoma five days following surgery and who give informed consent to enter the study will be randomized into two groups. Group A will be patients treated with a pressure dressing and observation, which is the most common current method of treatment. Group B will be patients treated with a VAC negative pressure device. Patients will be carefully monitored for continued drainage by evaluating the wounds and dressings clinically. Patients in either group that are still draining at ten days following surgery will be taken to the operating room for irrigation and debridement. Patients in either group who develop infection will be immediately treated with irrigation and debridement.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has had an orthopaedic surgical procedure following trauma and has a draining wound for at least five days
* No clinical evidence of infection
* Adult patient (19 years and older)

Exclusion Criteria:

* An infected hematoma. Infection will be defined by clinical signs and symptoms of infection that include increasing drainage, increasing pain, purulent drainage, and increasing erythema. Any hematomas that are thought to be infected will be cultured to confirm the diagnosis
* A surgical incision that can not be covered with VAC sponges and a water impermeable sheet (such Tegaderm) to achieve a closed vacuum environment over the wound
* Wounds associated with the surgical incision that are intentionally left open to heal with either a delayed primary closure or secondary granulation
* Abnormal coagulation leading to an expanding hematoma that will require surgical debridements
* Prisoners
* Pregnant Women
* Inability to comply with protocol
* Patients or family members who are unable or unwilling to sign study consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2001-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Dry and healed draining hematoma | If hematoma still draining 5 days post surgery, enter study; Still draining 10 days post surgery, return to OR for I&D

SECONDARY OUTCOMES:
Prevent development of infection | 5 - 10 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: David A Volgas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Ferdinando E, Guerin L, Jervis AO, Obidigbo H. Negative-pressure wound therapy and external fixation for infection and hematoma after hallux abducto valgus surgery. J Am Podiatr Med Assoc. 2007 Sep-Oct;97(5):410-4. doi: 10.7547/0970410. PMID 17901348